CLINICAL TRIAL: NCT06416527
Title: Effects of Pompage Associated or Not With Photobiomodulation on Pain, Range of Motion, and Quality of Life in Patients With Neck Pain: a Controlled, Randomized, and Double Blinded Study
Brief Title: Pompage and Photobiomodulation on Pain, Range of Motion, and Quality of Life in Patients With Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77505024300005511
Record Dates: First submitted 2024-04-30; First posted 2024-05-16 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-09

CONDITIONS: Cervicalgia
Keywords: neck pain; photobiomodulation; LED; manual therapy
MeSH Terms: conditions — Neck Pain | interventions — Low-Level Light Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: The participants will be divided into 2 groups:
  1. Pompage Group (Control): Patients will receive treatment through the application of the pompage technique in the cervical region during 10 sessions performed 3 times per week, excluding weekends.
  2. Pompage + FBM Group (Experimental): Treatment will consist of 10 sessions in which the pompage technique will be applied associated with photobiomodulation in the form of LED cluster in the cervical region, performed 3 times per week, excluding weekends.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study will be conducted by a team of researchers, including one researcher who will supervise the interventions, i.e., the application of pompages associated or not with PBM using LED clusters. This researcher will be the only one to know the intervention performed on each participant. Another researcher will conduct the initial assessment of outcomes and reevaluations (blinded to the experimental and control groups). The statistical analysis will also be performed blindly by a statistician who will receive the data without identification of the group. The patient will be blinded to the treatment with PBM (or its simulation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pompage and photobiomodulation (placebo) (Placebo Comparator): (1) Pompage Group + photobiomodulation placebo (Control): Patients will receive treatment through the application of the pompage technique in the cervical region during 10 sessions performed 3 times per week, excluding weekends.
  Interventions: Procedure: Pompage Technique (manual therapy); Device: Photobiomodulation (Placebo)
- Pompage + photobiomodulation (Experimental) (Experimental): (2) Pompage + photobiomodulation (PBM) Group (Experimental): Treatment will consist of 10 sessions in which the pompage technique will be applied associated with photobiomodulation in the form of LED cluster in the cervical region, performed 3 times per week, excluding weekends.
  Interventions: Device: Photobiomodulation (Experimental); Procedure: Pompage Technique (manual therapy)

INTERVENTIONS:
Device: Photobiomodulation (Experimental) — The photobiomodulation with a diode emitting light (LED) cluster device will be positioned on the cervical region of each patient (for 10 minutes each).
  Arms: Pompage + photobiomodulation (Experimental)
Procedure: Pompage Technique (manual therapy) — To perform cervical Pompage the patient lies comfortably on their back or sits upright. The therapist locates the target area on the cervical spine. Using gentle pressure, the therapist applies traction to the cervical spine, stretching the muscles and fascia. The traction is held for 20 seconds. The therapist then releases the traction, allowing the cervical spine to return to its neutral position. This process will be repeated 3 times, with adjustments made based on the patient's response and comfort level.
Device: Photobiomodulation (Placebo) — The photobiomodulation with a diode emitting light (LED) cluster device will be positioned on the cervical region of each patient (for 10 minutes each) with the device turned off (inactive), simulating the time with a recorded beep sound.
  Arms: Pompage and photobiomodulation (placebo)

SUMMARY:
The aim of this study is to evaluate the effects of Pompage associated or not with PBM, using a cluster of LEDs, on pain and neck disability. This controlled, randomized, and double-blinded clinical study includes participants of both genders, aged 18 to 55, with non-specific chronic neck pain will be included. Participants will be randomized into two groups: (1) Pompage (n=28) focusing only on manual therapy through Pompage technique and (2) Pompage + PBM Group (n=28) involving the same procedures as the first group, followed by PBM with a LED cluster applied for 10 minutes to the neck region for 10 sessions. Pain and functional disability will be assessed using the visual analog scale (VAS) and Neck Pain Disability Index before and after the intervention. The resulting data will be submitted to statistical analysis considering α=0.05.

DETAILED DESCRIPTION:
Chronic neck pain is a persistent condition affecting the spinal region, resulting in pain and restricted mobility. The management of neck pain often involves manual therapies, encompassing both passive and active interventions, aimed at alleviating pain, enhancing function, improving mobility, motor control, and reducing inflammatory processes. This pain can persist for at least three months and is considered non-specific when it is not associated with any specific underlying condition, such as inflammatory rheumatic disease, osteoporosis, cancer, or radiculopathy.

The use of lasers and LEDs for photobiomodulation (PBM) represents an advantageous approach to treating neck pain, given their demonstrated therapeutic efficacy in the literature. Moreover, these resources are non-invasive and easy to apply, making them an attractive option for both patients and healthcare professionals. Therefore, the aim of this study is to evaluate the effects of Pompage associated or not with PBM, using a cluster of LEDs, on pain and neck disability. This controlled, randomized, and double-blinded clinical study includes participants of both genders, aged 18 to 62, with non-specific chronic neck pain will be included. Participants will be randomized into two groups: (1) Pompage (n=28) focusing only on manual therapy through Pompage technique and (2) Pompage + PBM Group (n=28) involving the same procedures as the first group, followed by PBM with a LED cluster applied for 10 minutes to the neck region. The treatment protocol consists of 10 sessions, three times weekly, excluding weekends. For PBM, a cluster comprising 264 LEDs (8 mW; 4.89J; 9.6 J/cm2; 16 mW/cm² per LED) will be used, with 132 red (660nm) and 132 infrared (850nm) LEDs. Pain and functional disability will be assessed using the visual analog scale (VAS) and Neck Pain Disability Index before and after the intervention. The resulting data will be submitted to statistical analysis considering α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 62 years;
* Both genders;
* Without comorbidities.

Exclusion Criteria:

* Presentation of rheumatic or degenerative diseases in the cervical region;
* Undergoing orthodontic or physiotherapeutic treatment;
* Initiation of the use of any medication during any phase of the study;
* Using bite plate.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Pain baseline | Baseline
  The Visual Analog Scale (VAS) consists of a visual graduated scale from 0 to 10 cm, where 0 represents the absence of pain and 10 represents very intense pain, used to measure the pain experienced by the patient. This scale will be used for assessment and to monitor treatment progression. The patient is asked about the intensity of their pain, and the corresponding number on the scale is marked.
Pain at the end | At the 50th day of the protocol (at the end of Session 10)
  The Visual Analog Scale (VAS) consists of a visual graduated scale from 0 to 10 cm, where 0 represents the absence of pain and 10 represents very intense pain, used to measure the pain experienced by the patient. This scale will be used for assessment and to monitor treatment progression. The patient is asked about the intensity of their pain, and the corresponding number on the scale is marked.

SECONDARY OUTCOMES:
Cervical Range of Motion at baseline | Baseline
  The Goniometer is an instrument used to measure the degrees of range of motion (ROM) of the cervical region, with normal standards considered as follows: flexion from 0 to 65 degrees; extension from 0 to 50 degrees; lateral flexion to the right and left from 0 to 40 degrees; right and left rotation from 0 to 55 degrees. It will be used for assessment and monitoring of treatment progression.
Cervical Range of Motion at the end | At the 50th day of the protocol (at the end of Session 10)
  The Goniometer is an instrument used to measure the degrees of range of motion (ROM) of the cervical region, with normal standards considered as follows: flexion from 0 to 65 degrees; extension from 0 to 50 degrees; lateral flexion to the right and left from 0 to 40 degrees; right and left rotation from 0 to 55 degrees. It will be used for assessment and monitoring of treatment progression.
Quality of Life at baseline | Baseline
  To assess the quality of life of the participants, the WHOQOL-BREF will be utilized, an abbreviated instrument developed by the World Health Organization. This questionnaire will consist of 26 items distributed across four main domains: Physical, Psychological, Social Relationships, and Environment. Each item will be rated on a 5-point Likert scale, ranging from 1 ("not at all") to 5 ("extremely"). The scores for each domain will be calculated from the averages of the corresponding item responses, multiplied by 4 to transform the results into a scale of 0 to 100. Higher scores will indicate a better perception of quality of life in the specific domain
Quality of Life at the end | At the 50th day of the protocol (at the end of Session 10)
  To assess the quality of life of the participants, the WHOQOL-BREF will be utilized, an abbreviated instrument developed by the World Health Organization. This questionnaire will consist of 26 items distributed across four main domains: Physical, Psychological, Social Relationships, and Environment. Each item will be rated on a 5-point Likert scale, ranging from 1 ("not at all") to 5 ("extremely"). The scores for each domain will be calculated from the averages of the corresponding item responses, multiplied by 4 to transform the results into a scale of 0 to 100. Higher scores will indicate a better perception of quality of life in the specific domain
Degree of Functional Disability at the baseline | Baseline
  The Neck Disability Index (NDI) questionnaire, which assesses the degree of functional disability of the cervical region, is a self-administered questionnaire consisting of 10 sessions with 6 responses, reflecting 6 stages of functional disability, with scores ranging from 0 to 5, where 0 represents the lowest and 5 represents the highest level of disability.
Degree of Functional Disability at the end | At the 50th day of the protocol (at the end of Session 10)
  The Neck Disability Index (NDI) questionnaire, which assesses the degree of functional disability of the cervical region, is a self-administered questionnaire consisting of 10 sessions with 6 responses, reflecting 6 stages of functional disability, with scores ranging from 0 to 5, where 0 represents the lowest and 5 represents the highest level of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- UNINOVE, São Paulo, São Paulo, Brazil